CLINICAL TRIAL: NCT00157599
Title: A Cohort Study Evaluating the Safety of a Diagnostic Strategy Involving D-Dimer and Compression Ultrasonography in Patients With Suspected Recurrent Deep Vein Thrombosis
Brief Title: MDA D-Dimer / Recurrent DVT Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTMG-2002-MDA
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2007-10

CONDITIONS: Deep Vein Thrombosis
Keywords: deep vein thrombosis; DVT
MeSH Terms: conditions — Venous Thrombosis | interventions — cupric sulfide

INTERVENTIONS:
Procedure: various diagnostic measures for DVT (e.g., CUS)

SUMMARY:
To determine whether treatment and further investigation can be safely withheld in patients who present with suspected recurrent deep vein thrombosis (DVT) and have either a (i) negative D-Dimer or (ii) a positive D-Dimer with normal serial compression ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Currently suspected for recurrent DVT
* Has a prior history of objectively documented DVT or PE

Exclusion Criteria:

* Comorbid condition limiting survival to less than 3 months
* History of hypersensitivity to contrast medium
* Renal dysfunction with a creatinine of > 150 mcmol/L
* Treatment with full-dose therapeutic unfractionated or low molecular weight heparin that was initiated 24 hours or more prior to eligibility assessment
* Pregnancy or lactation
* Symptomatic for pulmonary embolism
* Absence of symptoms within five days prior to presentation
* Participation in another trial precluding the use of the diagnostic algorithm in this study
* Geographically inaccessible for follow-up
* Compression ultrasound, venogram, IPG, or D-dimer performed PRIOR to assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2002-01; Study Completion 2007-03

PRIMARY OUTCOMES:
Suspected DVT during follow-up
Suspected PE during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Bates, M.D., Principal Investigator — McMaster University
Locations (6):
- Canada (5):
  - Hamilton General Hospital, Hamilton, Ontario
  - McMaster University Medical Centre, Hamilton, Ontario
  - St. Joseph's Hospital, Hamilton, Ontario
  - Henderson Research Centre, Hamilton, Ontario
  - Sir Mortimer B. Davis Jewish General, Montreal, Quebec
- Academic Medical Centre, Amsterdam, Netherlands